CLINICAL TRIAL: NCT00001678
Title: Genetics of Rheumatoid Arthritis: The North American Rheumatoid Arthritis Consortium
Brief Title: Genetics of Rheumatoid Arthritis
Status: Completed | Type: Observational
Sponsor: National Institute of Arthritis and Musculoskeletal and Skin Diseases (NIAMS) (NIH)
Collaborators: National Human Genome Research Institute (NHGRI) (NIH)
Organization: National Institutes of Health Clinical Center (CC) (NIH)
Other Study IDs: 980124; 98-HG-0124
Record Dates: First submitted 1999-11-03; First posted 1999-11-04 (Estimated); Last update posted 2017-10-06 (Actual); Status verified 2014-06-20

CONDITIONS: Rheumatoid Arthritis
Keywords: Autoimmunity; Sibling Pairs; Genes; Rheumatoid Arthritis; Bone Erosion
MeSH Terms: conditions — Arthritis, Rheumatoid; Autoimmune Diseases

SUMMARY:
This study attempts to identify the genes responsible for rheumatoid arthritis (RA), or inflammation of the joints. It is known that genes play an important role in RA, but their number and significance have not been determined. RA tends to run in families. This study will examine the DNA (hereditary material) of patients with RA and their family members to try to determine which chromosomes(s) contain the genes responsible for the disease.

Patients with rheumatoid arthritis and their family members may be eligible for this study.

Participants with RA who have a brother or sister with RA will undergo the following procedures:

* Review of their medical records
* Medical history
* Examination of the joints
* Hand X-rays
* Blood tests

Participants who 1) do not have RA but who have a relative with the disease, or 2) have RA and a relative other than a brother or sister who has the disease will provide a blood sample or a buccal (cheek) cell sample. Cheek cells are obtained by swishing a small amount of mouthwash in the mouth or by lightly bushing the inside of the cheek with a swab or brush.

The samples will be tested for rheumatoid factor, DNA studies, and HLA type (a blood type found on white blood cells). Certain HLA types have been associated with an increased risk or severity of RA.

DETAILED DESCRIPTION:
The purpose of this protocol is to identify genetic susceptibility loci for rheumatoid arthritis. The Genetics and Genomics Branch of the Intramural Research Program of NIAMS [now the

Inflammatory Diseases Section of the Intramural Research Program of NHGRI] has joined with

several extramural centers to form the North American Rheumatoid Arthritis Consortium

(NARAC). The Consortium intends to identify and obtain clinical specimens on a total of 1000

sibling pairs with rheumatoid arthritis; up to 100 sibling pairs will be recruited at the Clinical

Center. Samples from parents and other family members will also be obtained, where

appropriate. Rheumatoid factors, HLA-DR typings, and hand films will be obtained on all

sibling pairs. In addition, DNA will be extracted from peripheral blood or buccal scrapings. The

DNA from all 1000 sibling pairs will be typed for a set of approximately 350 genetic markers in

order to identify chromosomal regions likely to harbor genes conferring susceptibility to

rheumatoid arthritis. For those chromosomal regions that are positive in this initial screen,

families will be genotyped for additional markers to define disease-associated haplotypes, and high density single nucleotide polymorphism (SNP) analysis will be conducted to narrow the regions of interest. Candidate genes will be chosen from the narrowed regions of interest, and/or based on functional considerations, and will be screened for mutations in rheumatoid arthritis.

ELIGIBILITY:
* INCLUSION CRITERIA:

SIBLING PAIR:

A diagnosis of rheumatoid arthritis in both sibs by the 1987 ACR criteria.

Definite bony erosions in at least one affected sibling.

Age of disease onset greater than 18 years and less than 60 years in at least one sibling.

Neither sibling has psoriasis, inflammatory bowel disease, or systemic lupus erythematosus.

BLOOD RELATIVES OF AFFECTED SIBLING PAIRS:

Age greater than 18 years.

Where possible, all other affected siblings will be invited to participate.

Where possible, both parents of affected siblings will be invited to participate.

Other relatives, both affected and unaffected, may be invited to participate if, in the opinion of the investigators, samples from these individuals would contribute important genetic information. Two cases in which this might happen are: a) extended families in which there are several affected individuals, where conventional linkage analysis might be applied; b) affected sibling pairs for which parents are unavailable, where additional siblings will provide information on parental alleles not transmitted to the affected siblings.

EXCLUSION CRITERIA FOR AFFECTED SIBLINGS:

Psoriasis, inflammatory bowel disease, systemic lupus erythematosus.

Inability to provide infomed consent.

The sole criterion for exclusion of adult blood relatives of affected sibling pairs would be inability to provide informed consent.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 39 (Actual)
Dates: Start 1998-07-07; Study Completion 2014-06-20

CONTACTS AND LOCATIONS:
Overall Officials: Daniel L Kastner, M.D., Principal Investigator — National Human Genome Research Institute (NHGRI)
Locations (1):
- National Institutes of Health Clinical Center, 9000 Rockville Pike, Bethesda, Maryland, United States

REFERENCES:
- [Background] Stastny P. Association of the B-cell alloantigen DRw4 with rheumatoid arthritis. N Engl J Med. 1978 Apr 20;298(16):869-71. doi: 10.1056/NEJM197804202981602. PMID 147420
- [Background] Lawrence RC, Hochberg MC, Kelsey JL, McDuffie FC, Medsger TA Jr, Felts WR, Shulman LE. Estimates of the prevalence of selected arthritic and musculoskeletal diseases in the United States. J Rheumatol. 1989 Apr;16(4):427-41. PMID 2746583
- [Background] Harris ED Jr. Rheumatoid arthritis. Pathophysiology and implications for therapy. N Engl J Med. 1990 May 3;322(18):1277-89. doi: 10.1056/NEJM199005033221805. No abstract available. PMID 2271017